CLINICAL TRIAL: NCT01061567
Title: Assessment of the Safety and Efficacy of Pramipexole Extended Release in Patients With Parkinson's Disease in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.675
Record Dates: First submitted 2009-12-24; First posted 2010-02-03 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Male and female patients with Parkinson's disease

SUMMARY:
The general aim of this non-interventional study is to assess the safety and efficacy of pramipexole extended release in patients with Parkinson's disease in routine clinical practice.

ELIGIBILITY:
Inclusion criteria:

* Early and advanced idiopathic Parkinson's disease
* Male and female patients over 18 years of age
* Indication for treatment with pramipexole ER according to Summary of Product Characteristics (SmPC)

Exclusion criteria:

* Ongoing treatment with pramipexole ER
* Exclusion criteria in line with the pramipexole ER SmPC:

In particular hypersensitivity to pramipexole or to any of the excipients and pregnancy and lactation as stated in the SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Probability Sample
Enrollment: 1814 (Actual)
Dates: Start 2009-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (284):
- Austria (111):
  - Boehringer Ingelheim Investigational Site 1, Bad Ischl
  - Boehringer Ingelheim Investigational Site 2, Bad Radkersburg
  - Boehringer Ingelheim Investigational Site 3, Baden
  - Boehringer Ingelheim Investigational Site 4, Baden
  - Boehringer Ingelheim Investigational Site 5, Bludenz
  - Boehringer Ingelheim Investigational Site 6, Braunau/Inn
  - Boehringer Ingelheim Investigational Site 7, Deutschlandsberg
  - Boehringer Ingelheim Investigational Site 8, Dornbirn
  - Boehringer Ingelheim Investigational Site 9, Dornbirn
  - Boehringer Ingelheim Investigational Site 10, Ehenbichl
  - Boehringer Ingelheim Investigational Site 11, Eisenstadt
  - Boehringer Ingelheim Investigational Site 12, Eisenstadt
  - Boehringer Ingelheim Investigational Site 13, Feldbach
  - Boehringer Ingelheim Investigational Site 14, Feldkirchen in Kärnten
  - Boehringer Ingelheim Investigational Site 15, Gänserndorf
  - Boehringer Ingelheim Investigational Site 16, Graz
  - Boehringer Ingelheim Investigational Site 17, Graz
  - Boehringer Ingelheim Investigational Site 18, Graz
  - Boehringer Ingelheim Investigational Site 19, Graz
  - Boehringer Ingelheim Investigational Site 20, Grieskirchen
  - Boehringer Ingelheim Investigational Site 21, Grimmenstein
  - Boehringer Ingelheim Investigational Site 22, Hainburg an der Donau
  - Boehringer Ingelheim Investigational Site 23, Hall/Tirol
  - Boehringer Ingelheim Investigational Site 24, Hallein
  - Boehringer Ingelheim Investigational Site 25, Hartberg
  - Boehringer Ingelheim Investigational Site 26, Hermagor
  - Boehringer Ingelheim Investigational Site 27, Hohenems
  - Boehringer Ingelheim Investigational Site 28, Horn
  - Boehringer Ingelheim Investigational Site 29, Horn
  - Boehringer Ingelheim Investigational Site 30, Imst
  - Boehringer Ingelheim Investigational Site 31, Innsbruck
  - Boehringer Ingelheim Investigational Site 32, Innsbruck
  - Boehringer Ingelheim Investigational Site 33, Innsbruck
  - Boehringer Ingelheim Investigational Site 34, Judenburg
  - Boehringer Ingelheim Investigational Site 35, Kapfenberg
  - Boehringer Ingelheim Investigational Site 36, Klagenfurt
  - Boehringer Ingelheim Investigational Site 37, Klagenfurt
  - Boehringer Ingelheim Investigational Site 38, Klagenfurt
  - Boehringer Ingelheim Investigational Site 39, Klagenfurt
  - Boehringer Ingelheim Investigational Site 40, Knittelfeld
  - Boehringer Ingelheim Investigational Site 41, Krems
  - Boehringer Ingelheim Investigational Site 42, Kufstein
  - Boehringer Ingelheim Investigational Site 43, Lassnitzhöhe
  - Boehringer Ingelheim Investigational Site 44, Leibnitz, Styria
  - Boehringer Ingelheim Investigational Site 45, Leoben
  - Boehringer Ingelheim Investigational Site 46, Lienz
  - Boehringer Ingelheim Investigational Site 47, Lienz
  - Boehringer Ingelheim Investigational Site 48, Lilienfeld
  - Boehringer Ingelheim Investigational Site 49, Linz
  - Boehringer Ingelheim Investigational Site 50, Linz
  - Boehringer Ingelheim Investigational Site 51, Melk
  - Boehringer Ingelheim Investigational Site 52, Mürzzuschlag
  - Boehringer Ingelheim Investigational Site 53, Neulengbach
  - Boehringer Ingelheim Investigational Site 54, Neulengbach
  - Boehringer Ingelheim Investigational Site 55, Neunkirchen
  - Boehringer Ingelheim Investigational Site 56, Neunkirchen
  - Boehringer Ingelheim Investigational Site 57, Neusiedl am See
  - Boehringer Ingelheim Investigational Site 58, Oberwart
  - Boehringer Ingelheim Investigational Site 59, Oberwart
  - Boehringer Ingelheim Investigational Site 60, Oberwart
  - Boehringer Ingelheim Investigational Site 61, Regelsbrunn
  - Boehringer Ingelheim Investigational Site 62, Ried im Innkreis
  - Boehringer Ingelheim Investigational Site 63, Ried im Innkreis
  - Boehringer Ingelheim Investigational Site 64, Rohrbach
  - Boehringer Ingelheim Investigational Site 65, Salzburg
  - Boehringer Ingelheim Investigational Site 66, Salzburg
  - Boehringer Ingelheim Investigational Site 67, Salzburg
  - Boehringer Ingelheim Investigational Site 68, Salzburg
  - Boehringer Ingelheim Investigational Site 71, Sankt Pölten
  - Boehringer Ingelheim Investigational Site 72, Sankt Pölten
  - Boehringer Ingelheim Investigational Site 73, Sankt Veit an der Glan
  - Boehringer Ingelheim Investigational Site 69, Scheibbs
  - Boehringer Ingelheim Investigational Site 70, St Johann im Pongau
  - Boehringer Ingelheim Investigational Site 74, Telfs
  - Boehringer Ingelheim Investigational Site 75, Tulln
  - Boehringer Ingelheim Investigational Site 76, Tullnerbach-Lawies
  - Boehringer Ingelheim Investigational Site 100, Vienna
  - Boehringer Ingelheim Investigational Site 101, Vienna
  - Boehringer Ingelheim Investigational Site 102, Vienna
  - Boehringer Ingelheim Investigational Site 103, Vienna
  - Boehringer Ingelheim Investigational Site 104, Vienna
  - Boehringer Ingelheim Investigational Site 105, Vienna
  - Boehringer Ingelheim Investigational Site 106, Vienna
  - Boehringer Ingelheim Investigational Site 107, Vienna
  - Boehringer Ingelheim Investigational Site 84, Vienna
  - Boehringer Ingelheim Investigational Site 85, Vienna
  - Boehringer Ingelheim Investigational Site 86, Vienna
  - Boehringer Ingelheim Investigational Site 87, Vienna
  - Boehringer Ingelheim Investigational Site 88, Vienna
  - Boehringer Ingelheim Investigational Site 89, Vienna
  - Boehringer Ingelheim Investigational Site 90, Vienna
  - Boehringer Ingelheim Investigational Site 91, Vienna
  - Boehringer Ingelheim Investigational Site 92, Vienna
  - Boehringer Ingelheim Investigational Site 93, Vienna
  - Boehringer Ingelheim Investigational Site 94, Vienna
  - Boehringer Ingelheim Investigational Site 95, Vienna
  - Boehringer Ingelheim Investigational Site 96, Vienna
  - Boehringer Ingelheim Investigational Site 97, Vienna
  - Boehringer Ingelheim Investigational Site 98, Vienna
  - Boehringer Ingelheim Investigational Site 99, Vienna
  - Boehringer Ingelheim Investigational Site 77, Villach
  - Boehringer Ingelheim Investigational Site 78, Villach
  - Boehringer Ingelheim Investigational Site 79, Villach-Warmbad
  - Boehringer Ingelheim Investigational Site 80, Vöcklabruck
  - Boehringer Ingelheim Investigational Site 81, Vöcklabruck
  - Boehringer Ingelheim Investigational Site 82, Völkermarkt
  - Boehringer Ingelheim Investigational Site 83, Wagna
  - Boehringer Ingelheim Investigational Site 108, Wiener Neustadt
  - Boehringer Ingelheim Investigational Site 109, Wolfsberg
  - Boehringer Ingelheim Investigational Site 110, Zirl
  - Boehringer Ingelheim Investigational Site 111, Zwettl Stadt
- Estonia (10):
  - Boehringer Ingelheim Investigational Site 115, Järvamaa
  - Boehringer Ingelheim Investigational Site 114, Kohtla-Järve
  - Boehringer Ingelheim Investigational Site 121, Kuressaare
  - Boehringer Ingelheim Investigational Site 116, Rakvere
  - Boehringer Ingelheim Investigational Site 112, Tallinn
  - Boehringer Ingelheim Investigational Site 113, Tallinn
  - Boehringer Ingelheim Investigational Site 117, Tartu
  - Boehringer Ingelheim Investigational Site 118, Valga
  - Boehringer Ingelheim Investigational Site 119, Viimsi
  - Boehringer Ingelheim Investigational Site 120, Viljandi
- Kazakhstan (3):
  - Boehringer Ingelheim Investigational Site 283, Almaty
  - Boehringer Ingelheim Investigational Site 284, Astana
  - Boehringer Ingelheim Investigational Site 282, Shymkent
- Romania (82):
  - Boehringer Ingelheim Investigational Site 193, Alba Iulia
  - Boehringer Ingelheim Investigational Site 194, Bacau
  - Boehringer Ingelheim Investigational Site 195, Bacau
  - Boehringer Ingelheim Investigational Site 196, Bacau
  - Boehringer Ingelheim Investigational Site 197, Baia Mare
  - Boehringer Ingelheim Investigational Site 198, Baia Mare
  - Boehringer Ingelheim Investigational Site 199, Botoșani
  - Boehringer Ingelheim Investigational Site 200, Brasov
  - Boehringer Ingelheim Investigational Site 201, Brasov
  - Boehringer Ingelheim Investigational Site 202, Bucharest
  - Boehringer Ingelheim Investigational Site 203, Bucharest
  - Boehringer Ingelheim Investigational Site 204, Bucharest
  - Boehringer Ingelheim Investigational Site 205, Bucharest
  - Boehringer Ingelheim Investigational Site 206, Bucharest
  - Boehringer Ingelheim Investigational Site 207, Bucharest
  - Boehringer Ingelheim Investigational Site 208, Bucharest
  - Boehringer Ingelheim Investigational Site 209, Bucharest
  - Boehringer Ingelheim Investigational Site 210, Bucharest
  - Boehringer Ingelheim Investigational Site 211, Bucharest
  - Boehringer Ingelheim Investigational Site 212, Bucharest
  - Boehringer Ingelheim Investigational Site 213, Bucharest
  - Boehringer Ingelheim Investigational Site 214, Bucharest
  - Boehringer Ingelheim Investigational Site 215, Bucharest
  - Boehringer Ingelheim Investigational Site 216, Bucharest
  - Boehringer Ingelheim Investigational Site 217, Bucharest
  - Boehringer Ingelheim Investigational Site 218, Bucharest
  - Boehringer Ingelheim Investigational Site 219, Bucharest
  - Boehringer Ingelheim Investigational Site 220, Buzău
  - Boehringer Ingelheim Investigational Site 221, Buzău
  - Boehringer Ingelheim Investigational Site 222, Campulung Muscel
  - Boehringer Ingelheim Investigational Site 223, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 224, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 225, Constanța
  - Boehringer Ingelheim Investigational Site 226, Constanța
  - Boehringer Ingelheim Investigational Site 227, Constanța
  - Boehringer Ingelheim Investigational Site 228, Craiova
  - Boehringer Ingelheim Investigational Site 229, Craiova
  - Boehringer Ingelheim Investigational Site 230, Craiova
  - Boehringer Ingelheim Investigational Site 231, Craiova
  - Boehringer Ingelheim Investigational Site 232, Craiova
  - Boehringer Ingelheim Investigational Site 233, Curtea de Argeş
  - Boehringer Ingelheim Investigational Site 234, Focşani
  - Boehringer Ingelheim Investigational Site 235, Focşani
  - Boehringer Ingelheim Investigational Site 236, Galati
  - Boehringer Ingelheim Investigational Site 237, Iași
  - Boehringer Ingelheim Investigational Site 238, Iași
  - Boehringer Ingelheim Investigational Site 239, Iași
  - Boehringer Ingelheim Investigational Site 240, Medgidia
  - Boehringer Ingelheim Investigational Site 241, Oradea
  - Boehringer Ingelheim Investigational Site 242, Oradea
  - Boehringer Ingelheim Investigational Site 243, Piatra Neamţ
  - Boehringer Ingelheim Investigational Site 244, Piatra Neamţ
  - Boehringer Ingelheim Investigational Site 245, Piteşti
  - Boehringer Ingelheim Investigational Site 246, Piteşti
  - Boehringer Ingelheim Investigational Site 247, Ploieşti
  - Boehringer Ingelheim Investigational Site 248, Prahova
  - Boehringer Ingelheim Investigational Site 249, Radauti
  - Boehringer Ingelheim Investigational Site 250, Râmnicu Vâlcea
  - Boehringer Ingelheim Investigational Site 251, Râmnicu Vâlcea
  - Boehringer Ingelheim Investigational Site 252, Râmnicu Vâlcea
  - Boehringer Ingelheim Investigational Site 253, Satu Mare
  - Boehringer Ingelheim Investigational Site 254, Satu Mare
  - Boehringer Ingelheim Investigational Site 255, Sibiu
  - Boehringer Ingelheim Investigational Site 256, Sibiu
  - Boehringer Ingelheim Investigational Site 257, Simleul Silvaniei
  - Boehringer Ingelheim Investigational Site 258, Slobozia
  - Boehringer Ingelheim Investigational Site 259, Suceava
  - Boehringer Ingelheim Investigational Site 260, Târgovişte
  - Boehringer Ingelheim Investigational Site 261, Târgovişte
  - Boehringer Ingelheim Investigational Site 262, Târgu Mureş
  - Boehringer Ingelheim Investigational Site 263, Târnăveni
  - Boehringer Ingelheim Investigational Site 264, Târnăveni
  - Boehringer Ingelheim Investigational Site 265, Timișoara
  - Boehringer Ingelheim Investigational Site 266, Timișoara
  - Boehringer Ingelheim Investigational Site 267, Timișoara
  - Boehringer Ingelheim Investigational Site 268, Timișoara
  - Boehringer Ingelheim Investigational Site 269, Tulcea
  - Boehringer Ingelheim Investigational Site 270, Tulcea
  - Boehringer Ingelheim Investigational Site 271, Tulcea
  - Boehringer Ingelheim Investigational Site 272, Turda
  - Boehringer Ingelheim Investigational Site 273, Turnu Măgurele
  - Boehringer Ingelheim Investigational Site 274, Zalău
- Serbia (7):
  - Boehringer Ingelheim Investigational Site 275, Belgrade
  - Boehringer Ingelheim Investigational Site 276, Belgrade
  - Boehringer Ingelheim Investigational Site 278, Kragujevac
  - Boehringer Ingelheim Investigational Site 281, Kraljevo
  - Boehringer Ingelheim Investigational Site 279, Niš
  - Boehringer Ingelheim Investigational Site 277, Novi Sad
  - Boehringer Ingelheim Investigational Site 280, Užice
- Slovakia (61):
  - Boehringer Ingelheim Investigational Site 122, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 123, Bardejov
  - Boehringer Ingelheim Investigational Site 124, Bardejov
  - Boehringer Ingelheim Investigational Site 125, Bratislava
  - Boehringer Ingelheim Investigational Site 126, Bratislava
  - Boehringer Ingelheim Investigational Site 127, Bratislava
  - Boehringer Ingelheim Investigational Site 128, Bratislava
  - Boehringer Ingelheim Investigational Site 129, Bratislava
  - Boehringer Ingelheim Investigational Site 130, Bratislava
  - Boehringer Ingelheim Investigational Site 131, Bratislava
  - Boehringer Ingelheim Investigational Site 132, Bratislava
  - Boehringer Ingelheim Investigational Site 133, Brezno
  - Boehringer Ingelheim Investigational Site 134, Detva
  - Boehringer Ingelheim Investigational Site 135, Dolný Kubín
  - Boehringer Ingelheim Investigational Site 136, Dolný Kubín
  - Boehringer Ingelheim Investigational Site 137, Hlohovec
  - Boehringer Ingelheim Investigational Site 138, Hlohovec
  - Boehringer Ingelheim Investigational Site 139, Humenné
  - Boehringer Ingelheim Investigational Site 140, Kežmarok
  - Boehringer Ingelheim Investigational Site 141, Kežmarok
  - Boehringer Ingelheim Investigational Site 142, Komárno
  - Boehringer Ingelheim Investigational Site 143, Košice
  - Boehringer Ingelheim Investigational Site 144, Košice
  - Boehringer Ingelheim Investigational Site 145, Košice
  - Boehringer Ingelheim Investigational Site 146, Košice
  - Boehringer Ingelheim Investigational Site 147, Košice
  - Boehringer Ingelheim Investigational Site 148, Krompachy
  - Boehringer Ingelheim Investigational Site 149, Liptovský Mikulás
  - Boehringer Ingelheim Investigational Site 150, Lučenec
  - Boehringer Ingelheim Investigational Site 151, Lučenec
  - Boehringer Ingelheim Investigational Site 152, Lučenec
  - Boehringer Ingelheim Investigational Site 153, Martin
  - Boehringer Ingelheim Investigational Site 154, Martin
  - Boehringer Ingelheim Investigational Site 155, Myjava
  - Boehringer Ingelheim Investigational Site 156, Námestovo
  - Boehringer Ingelheim Investigational Site 157, Nitra
  - Boehringer Ingelheim Investigational Site 158, Nitra
  - Boehringer Ingelheim Investigational Site 159, Nitra
  - Boehringer Ingelheim Investigational Site 160, Nitra
  - Boehringer Ingelheim Investigational Site 161, Pezinok
  - Boehringer Ingelheim Investigational Site 162, Piešťany
  - Boehringer Ingelheim Investigational Site 163, Prešov
  - Boehringer Ingelheim Investigational Site 164, Prešov
  - Boehringer Ingelheim Investigational Site 165, Prešov
  - Boehringer Ingelheim Investigational Site 166, Prešov
  - Boehringer Ingelheim Investigational Site 169, Skalica
  - Boehringer Ingelheim Investigational Site 170, Stará Lubovna
  - Boehringer Ingelheim Investigational Site 167, Šahy
  - Boehringer Ingelheim Investigational Site 168, Šaľa
  - Boehringer Ingelheim Investigational Site 171, Šurany
  - Boehringer Ingelheim Investigational Site 172, Topoľčany
  - Boehringer Ingelheim Investigational Site 173, Trebišov
  - Boehringer Ingelheim Investigational Site 174, Trencín
  - Boehringer Ingelheim Investigational Site 175, Trnava
  - Boehringer Ingelheim Investigational Site 176, Trnava
  - Boehringer Ingelheim Investigational Site 177, Trstená
  - Boehringer Ingelheim Investigational Site 178, Vranov Nad Top?ou
  - Boehringer Ingelheim Investigational Site 182, Zlaté Moravce
  - Boehringer Ingelheim Investigational Site 181, Zvolen
  - Boehringer Ingelheim Investigational Site 179, Žiar nad Hronom
  - Boehringer Ingelheim Investigational Site 180, Žilina
- Slovenia (10):
  - Boehringer Ingelheim Investigational Site 183, Celje
  - Boehringer Ingelheim Investigational Site 184, Lesce
  - Boehringer Ingelheim Investigational Site 185, Ljubljana
  - Boehringer Ingelheim Investigational Site 186, Ljubljana
  - Boehringer Ingelheim Investigational Site 187, Maribor
  - Boehringer Ingelheim Investigational Site 188, Maribor
  - Boehringer Ingelheim Investigational Site 190, Sempeter
  - Boehringer Ingelheim Investigational Site 191, Sempeter
  - Boehringer Ingelheim Investigational Site 189, Slovenj Gradec
  - Boehringer Ingelheim Investigational Site 192, Velenje

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Patients with Parkinson's disease in routine clinical practice.
Period: Overall Study
Arm/Group | All Patients
Started | 1814
Completed | 1738
Not Completed | 76
Not completed — Adverse Event | 32
Not completed — Death | 2
Not completed — Lack of Efficacy | 3
Not completed — Lost to Follow-up | 24
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 11
Not completed — Other reason than stated above | 3

BASELINE CHARACTERISTICS:
Population: Patients from Treated Set (TS) who were documented to have taken at least one dose of study treatment.
Arm/Group | All Patients
Number analyzed (Participants) | 1814
Age, Continuous [Mean (Standard Deviation); unit: years] — For 19 patients no data for age was documented, so the age was available for N=1795 patients
  years | 68.8 (9.2)
Gender [Number; unit: participants] — The documentation of gender was missing for 15 patients.
  participants
    Female | 910
    Male | 889

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: The number of patients with any adverse events (AEs), patients with drug-related AEs.
Time Frame: From the treatment initiation to the end of study, on average 92.9 days
Population: Patients from the Treated Set (TS).
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1814
participants
  Patients with any AE | 105
  Patients with drug-related AEs | 56

2. Primary Outcome: Proportion of Patients With Withdrawals Due to Adverse Events.
Description: Patients who discontinued treatment due to adverse events including deaths.
Time Frame: 16 weeks
Population: Patients from the Treated Set (TS).
Measure: Number; unit: proportion of participants
Arm/Group | All Patients
Number analyzed (Participants) | 1814
proportion of participants | 0.019

3. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Parts I and III Total Score
Description: Mentation, behaviour and mood is scored from 0-16 in UPDRS I (0 = best score to 16 = worst score), result of motor examination scored from 0-108 in UPDRS III (0=no disability, 108=maximum disability) . The change was calculated by Baseline value minus value at visit 3. A decrease (change>0) in the score means improvement.
Time Frame: Baseline and the end of study (up to 16 weeks)
Population: Patients from the Full Analysis Set (FAS) which includes all treated patients who have data for at least one post baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 1807
units on a scale
  UPDRS Part I score (N=1756) | 1.1 (1.6)
  UPDRS Part III score (N=1670) | 10.6 (9.4)

4. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Responder Rate
Description: The CGI-I was rated (from 1: very much improved, to 7: very much worse) to assess the overall status of Parkinson's disease. The clinician rated how much a patient's condition had improved or worsened relative to baseline state. The patients are considered to be a CGI-I responder if they are rated at least by minimally improved.
Time Frame: Baseline and the end of study (up to 16 weeks)
Population: Patients from FAS
Measure: Number; unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 1807
percentage of participants | 84.3

5. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) of Patient Satisfaction
Description: The visual analogue scale measures overall patient satisfaction with treatment on a continuous axis ranging from 0 (no satisfaction) to 100 (highest patient satisfaction). The change was calculated by the value at the final visit minus the value at baseline. Therefore, an increase (change>0) reflects an improvement in patient satisfaction.
Time Frame: Baseline and the end of study (up to 16 weeks)
Population: Patients from FAS with evaluable data in VAS at baseline and at visit 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 1657
units on a scale | 18.5 (22.6)

6. Secondary Outcome: Change From Baseline in Morisky Medication Adherence Scale (MMAS) 4 Item Score
Description: The Morisky Medication Adherence Scale with 4 items was administered to examine medication adherence. The score ranges from 0 (best adherence) to 4 (worst adherence). The change was calculated by the value at baseline minus the value at visit 3. Therefore, a change >0 reflects an improvement
Time Frame: Baseline and the end of study (up to 16 weeks)
Population: Patients from FAS with evaluable data in the Morisky scale for baseline and at visit 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 1629
units on a scale | 0.6 (1.1)

ADVERSE EVENTS:
Time Frame: From the treatment initiation to the end of study, on average 92.9 days
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 4/1814
Other Adverse Events (participants affected / at risk) | 0/1814
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=1814)
Cerebral insult (Nervous system disorders) | 1
Gambling (Psychiatric disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Heart failure (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
There was no PI assigned for the overall study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: Other
There was no PI assigned for the overall study